CLINICAL TRIAL: NCT01122147
Title: Phase 1 Evaluation of Therapeutic Effect of Chamomilla Tincture Mouthwash on Oral Aphthae
Brief Title: Clinical Evaluation of Fluid Extract of Chamomilla Tincture for Oral Aphthae
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Dental Research center of Mashhad Dental School, Mashhad University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 87034
Record Dates: First submitted 2010-05-07; First posted 2010-05-13 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2010-03

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Aphthous stomatitis; Herbal medicines; Matricaria Chamomilla
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- chamomilla tincture mouthwash (Active Comparator): Chamomile comprises bisaboloids, matricine and chamazulene, flavonoids, and cumarins having therapeutical anti-inflammatory, analgesic, musculotropic, and spasmolytic action
  Interventions: Drug: chamomilla tincture mouthwash
- placebo mouth wash (Placebo Comparator): placebo mouthwash is produced with the same taste and smell for using in placebo/ control group.
  Interventions: Drug: placebo mouthwash

INTERVENTIONS:
Drug: chamomilla tincture mouthwash — The patient is directed to mouth wash chamomilla tincture lightly three times a day,ten drops for each time,until ulcers completely heal
  Arms: chamomilla tincture mouthwash
Drug: placebo mouthwash — The patient is directed to use placebo mouthwash three times a day, ten drops for each time,until the ulcers completely heal
  Arms: placebo mouth wash

SUMMARY:
Recurrent aphthous stomatitis is a difficult to treat and quite common chronic inflammatory disease of the oral mucosa. This study evaluates the fluid extract from Chamomilla recutita's safety and effectiveness in treatment of aphthous stomatitis .

ELIGIBILITY:
Inclusion Criteria:• Confirmation of clinical diagnosis of aphthae

* Having the experience of oral aphthae at least once in a month
* Two weeks wash out periods after the last treatment

Exclusion Criteria:

* History of any systemic disease
* Using drugs which affect immune system
* Pregnancy and breast feeding
* Aphthous related syndromes

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
protocol designed to evaluate the effect of fluid extract from Chamomilla recutita's on treatment of aphthous stomatitis | 3 months
  This study evaluates the fluid extract from Chamomilla recutita's effectiveness on healing rate of aphthous stomatitis, and reducing ulcer size

SECONDARY OUTCOMES:
This study aimed to evaluate the efficacy of chamomile mouthwash of decreasing the pain and frequency of oral aphthous ulcer | 3 months
  In the present work the Analogical Visual Scale is used TO evaluate pain,and we also record the frequency of ulcers monthly

CONTACTS AND LOCATIONS:
Overall Officials: seyyed amir seyyedi, DDS-MSc, Principal Investigator — mashhad UMS
Locations (1):
- Mashhad University of Madical Science,Research Center of Mashhad Dental School, Mashhad, Khorasan Razavi, Iran